CLINICAL TRIAL: NCT00687258
Title: Evaluation Of The Impact Of A New Synthetic Vitamin E-Bonded Membrane On The Anemia And Oxidative Stress In End-Stage Renal Disease (ESRD) Patients
Brief Title: Evaluation Of A New Vitamin E-Bonded Membrane On Anemia And Oxidative Stress In End-Stage Renal Disease Patients
Acronym: Vi-E
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: A. Manzoni Hospital (Other)
Responsible Party: Principal Investigator, Simeone Andrulli, MD, Simeone Andrulli, MD, A. Manzoni Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vit E-Rif01-1
Record Dates: First submitted 2008-05-06; First posted 2008-05-30 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Anemia
Keywords: Anemia; Oxidative Stress; Erythropoietin; dialyser membrane; Vitamin E; Erythropoietin responsiveness; Erythropoietin resistance; hemodialysis
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): VitabranE ViE: Vitamin E-bonded polysulfone dialyzer
  Interventions: Device: VitabranE ViE
- 2 (No Intervention): APS-U (Asahi Polysulfone APS): Polysulfone dialyzer

INTERVENTIONS:
Device: VitabranE ViE — Polysulfone dialyser with vitamin E alpha-tocopherol
  Other Names: Vitamin E-bonded polysulfone dialyzer
  Arms: 1

SUMMARY:
The main purpose of this longitudinal study is to point out the effect of VitabranE on the ESA resistance and on the anemia observed in HD patients undergoing EPO maintenance therapy.

As a secondary purpose we will consider the effect of VitabranE on inflammation and oxidative stress parameters as a function of the changes observed in the anemia parameters.

DETAILED DESCRIPTION:
Aim

The aim of this pilot randomized study is to verify whether the addition of vitamin E alpha-tocopherol to the blood-side layer of a synthetic polysulfone dialyser membrane has a clinical advantage in terms of ESA responsiveness and, consequently, the anemic status of hemodialysed patients.

Patients

Patients of both genders aged more than 18 years will be considered eligible for the study if they had been receiving bicarbonate hemodialysis treatment for at least six months and stable ESA therapy for at least three months, and had adequate iron stores (ferritin levels >200 ng/ml and transferrin saturation >20%). Patients with haemoglobinopathies, sickle cell anemia, thalassemia or malignancies will be excluded, as were those who had experienced infection, vascular access thrombosis, stroke, myocardial infarction, heavy blood loss, major surgery or blood transfusion in the previous three months.

Study design

This is an 8-month, controlled and randomised study of two parallel groups; after giving their informed consent, the enrolled patients will be randomly assigned to the Vi-E experimental treatment (polysulfone dialyser with vitamin E alpha-tocopherol) or the PS control treatment (polysulfone dialyser without vitamin E alpha-tocopherol).

Clinical data

The dialyser will be randomly assigned at the beginning of the study, and pre and end-dialysis body weight, blood pressure and heart rate will be recorded at baseline and every two months. Dialysis prescription will not change during the study. All of the drugs administered during each dialysis session will be recorded, as all of the prescribed inter-dialysis therapies.

Laboratory data

Hemoglobin, serum albumin and plasma high-sensitivity C reactive protein levels (ELISA) will be recorded at baseline and every other month, together with nutritional and inflammation indices. Iron status will be evaluated on the basis of transferrin saturation and plasma ferritin levels. Reticulocytes and PTH levels will be also recorded. Equilibrated Kt/V will be calculated in order to estimate the dialysis dose of low molecular weight uraemic toxins, and the appearance of urea nitrogen will be calculated in order to estimate daily protein intake.

Plasma alpha-tocopherol and gamma tocopherol levels will be determined by means of reverse-phase HPLC analysis; total antioxidant capacity (TAC) will be determined using the ferric reducing-antioxidant power and advanced glycation end-products will be detected using total fluorescence at 335/385 Ex/Em. Advanced oxidation protein products, carbonyl products, erythrocyte creatine and interleukin 6 will be also determined.

Main response variable

The primary outcome measure will be the ESA resistance index, a combined variable calculated by dividing the weekly ESA dose by haemoglobin level and end-dialysis body weight.

Sample size

Given the pilot nature of the study, it is estimated that a sample of twenty patients (ten patients per group) will be sufficient to provide reasonable control over random variations in ESA resistance.

Statistical analysis

The data will be described using median values and interquartile ranges based on 25th and 75th percentiles for the distributed continuous variables. The baseline distribution of the continuous and categorical variables by group will be investigated using the Mann-Whitney and Chi-squared tests as appropriate.

The follow-up data will be analyzed using analysis of variance for repeated measures in order to test the possible differences in ESA resistance over time between the two groups.

A secondary analysis will be made by adding the values of some baseline covariates in order to identify predictors associated with ESA resistance. In order to reduce over-parameterizing the model, the explored covariates will be grouped in two hierarchical steps:

1. Biocompatibility of the previous membrane (categorical), iron status (transferrin saturation and ferritin), nutrition (albumin), intact PTH, inflammation (high- sensitivity C reactive protein);
2. Add some markers of oxidative stress (TAC, alpha- and gamma-TOC, carbonyl products, AOPP, AGEs and erythrocyte creatine) The effect of the experimental treatment over time will be tested by means of group interaction, with this hierarchical approach.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, aged ≥ 18, stabilized on BHD for at least 6 months.
2. Clinical stability during the last 3 months.
3. Serum Ferritin > 200 mg/L and Transferrin saturation >30%.
4. Maintenance therapy with epoetin alfa/beta or darbepoetin alfa.

Exclusion Criteria:

1. One of the following condition in the last 3 months :

   * acute infection
   * vascular access thrombosis
   * ictus cerebri
   * myocardial stroke
   * haemorrhage
   * major surgery
   * haemo-transfusion
2. Haemoglobinopaty, sickle cell anemia, familial erythroblastic anemia and any other haematological disorder interfering with the aim of the study
3. Malignancy
4. Participation to other studies or use of EPO analogues not yet commercialized
5. pharmacological dosage administration of antioxidant supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-07; Primary Completion 2007-03 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the ESA resistance index, a combined variable calculated by dividing the weekly ESA dose by haemoglobin level and end-dialysis body weight. | every other month

SECONDARY OUTCOMES:
Inflammatory status (CRP and IL-6) and oxidative stress markers (Vitamin E levels, TAC, Protein carbonyls and AOPP, AGEs). | every other month

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Locatelli, MD, Principal Investigator — Nephrology and Dialysis Department - A. Manzoni Hospital
Locations (1):
- Alessandro Manzoni Hospital, Nephrology and Dialysis Department, Lecco, Italy

REFERENCES:
- [Result] Andrulli S, Di Filippo S, Manzoni C, Stefanelli L, Floridi A, Galli F, Locatelli F. Effect of synthetic vitamin E-bonded membrane on responsiveness to erythropoiesis-stimulating agents in hemodialysis patients: a pilot study. Nephron Clin Pract. 2010;115(1):c82-9. doi: 10.1159/000294281. Epub 2010 Mar 8. PMID 20215781